CLINICAL TRIAL: NCT02587572
Title: A Randomized, Blinded and Placebo-controlled Trial to Evaluate the Safety and Efficacy of Allogeneic Human Mesenchymal Stem Cells in Patients With Metabolic Syndrome.
Brief Title: Safety and Efficacy Trial Using Allogeneic Human Mesenchymal Stem Cells: The SIRONA Trial
Acronym: SIRONA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor has made decision not to conduct this clinical trial.
Sponsor: Longeveron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-0000-02
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Metabolic Disease; Endothelial Dysfunction
MeSH Terms: conditions — Metabolic Diseases | interventions — Biological Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LMSCs 10 million IV (Experimental): A total of 10 subjects will receive: A single peripheral intravenous (IV) infusion of 10 x10^6 (10 million) of LMSCs to be administered on day 1.
  Interventions: Biological: Peripheral Intravenous (IV) infusion of LMSCs
- Placebo (Plasmalyte A,HSA) IV (Placebo Comparator): 10 subjects will receive: A single peripheral intravenous (IV) infusion of Plasmalyte A containing human serum albumin (HSA) to be administered on day 1.
  Interventions: Biological: Peripheral Intravenous (IV) infusion of LMSCs
- LMSCs 20 million IV (Experimental): 10 subjects will receive: A single peripheral intravenous (IV) infusion of 20x10^6 (20 million) LMSCs to be administered on day 1.
  Interventions: Biological: Peripheral Intravenous (IV) infusion of LMSCs
- LMSCs100 million IV (Experimental): 10 subjects will receive: A single peripheral intravenous (IV) infusion of 100x10^6 (100 million) LMSCs to be administered on day 1.
  Interventions: Biological: Peripheral Intravenous (IV) infusion of LMSCs

INTERVENTIONS:
Biological: Peripheral Intravenous (IV) infusion of LMSCs — Peripheral Intravenous (IV) infusion of LMSCs
  Other Names: LMSCs; Biological

SUMMARY:
This is a phase 2b, randomized, placebo-controlled clinical trial designed to evaluate the safety and efficacy of Longeveron Mesenchymal Stem Cells (LMSCs) in subjects with metabolic syndrome and to assess the effects of LMSCs on endothelial function using several different doses.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled clinical trial designed to evaluate the safety and efficacy of Longeveron Mesenchymal Stem Cells (LMSCs) in subjects with metabolic syndrome and to assess the effects of LMSCs on endothelial function using several different doses. Following a successful run-in phase, a total of forty (40) subjects will be randomized (1:1:1:1) to receive one of three different doses of LMSCs or placebo. After randomization, baseline imaging, testing and study product infusion, subjects will be followed up at 24 hours, month 1, month 3, month 6, month 9 and month 12 post study product infusion. All endpoints will be assessed at the 3, 6 and 12 month visits which will occur 90±30 days, 180±30 days, and 365±30 days respectively from the day of the study product infusion (Day 1). For the purposes of the endpoint analysis and safety evaluations, an "intent-to-treat" study population will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must provide written informed consent.
* Each subject must be ≥45 and ≤ 85 years of age at the time of signing the Informed Consent Form.
* Each subject must have endothelial dysfunction.
* At the time of enrollment, each subject must meet at least 3 out of the 5 criteria under the harmonized definition of the metabolic syndrome, consisting of the following

  * Hypertension.
  * Elevated triglycerides.
  * Reduced high-density lipoprotein (HDL) levels.
  * Elevated fasting glucose. --Central obesity.

Exclusion Criteria:

* Be unable and/or unwilling to perform any of the assessments required for endpoint analysis.
* Have diabetic retinopathy.
* Sitting or resting systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg at Screening.
* Have a resting blood oxygen saturation of <93% (measured by pulse oximetry).
* Be hypersensitive to dimethyl sulfoxide (DMSO).
* Have a history of alcohol or drug abuse within the past 24 months.
* Have been diagnosed with malignancy within the past 5 years, with the exception of curatively-treated basal cell carcinoma, melanoma in situ or cervical carcinoma.
* Be an organ transplant recipient.
* Be actively listed (or expected to be listed) for transplant of any organ.
* Have a condition that limits life expectancy to < 1 year.
* Be serum positive for HIV, hepatitis B sAG or viremic hepatitis C.
* Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraception (female patients must undergo a blood or urine pregnancy test at screening and within 36 hours prior to injection).
* Have any serious comorbid illness or other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.
* Be currently participating in an investigational therapeutic or device trial.
* Be currently participating in an investigational therapeutic or device trial, or have participated in an investigational therapeutic or device trial within the previous 30 days, or participate in any other clinical trial for the duration of the time that he or she is actively participating in this trial.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial function: Changes in endothelial function as assessed by the following: | 1 month post infusion
  Flow-mediated vasodilation (FMD). Endothelial progenitor cell (EPC) function.

SECONDARY OUTCOMES:
Difference in rate of change in the metabolic syndrome as defined by the following: | Baseline, 3 month, 6 month and 12 months.
  Endothelial function (FMD, EPC function) Inflammatory markers (CBC with differential, TNFα, CRP, IL-1, IL-6, D-dimer, Fibrinogen) Heart function and structure (Dobutamine Stress Echocardiography) Blood pressure Lipid profile (HDL; LDL; triglycerides; cholesterol) Physical activity (6 minute walk test and CHAMPS questionnaire) Lung function (spirometry) Glycemia (hemoglobin A1c;fasting glucose; urine glucose) Weight Subject quality of life (QOL) (QOL assessments).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Oliva, PhD, Study Director — Longeveron Inc.